CLINICAL TRIAL: NCT00963755
Title: Impact of F-18-Fluorocholine PET/CT and MR Imaging/ Spectroscopy in the Management of Primary and Recurrent Prostate Cancer
Brief Title: F-18-Fluorocholine PET/CT and MR Imaging/ Spectroscopy in the Management of Primary and Recurrent Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Principal Investigator, John O. Prior, Professor and Department Head, University of Lausanne Hospitals
Other Study IDs: 178/08
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
Keywords: Imaging; Positron emission tomography; F-18-FCH; Magnetic resonance imaging; Magnetic resonance spectroscopy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surgical specimen for total prostatectomy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary prostate cancer: Patients referred with a suspicion of prostate cancer based on elevated PSA and rectal examination in whom a prostate biopsy is planned and radical prostatectomy is envisioned in the event of a positive biopsy finding
- Prostate cancer relapse: Patients previously treated for prostate cancer and being investigated for biochemical relapse, (mostly in the Urology and Radiation Therapy Department, but not exclusively), for whom surgical or radiation therapy is envisioned in the event of a positive FCH-PET finding

SUMMARY:
The purpose of this study is to demonstrate that realization of guided biopsies by multimodal imaging with 18F-fluorocholine PET / CT and MR Imaging/spectroscopy would allow to increase the rate of detection prostate cancer compared with the current approach and give an information about location and tumoral volume before surgery.:

DETAILED DESCRIPTION:
1. To evaluate the utility of F-18-FCH-PET/CT and MR imaging with 3-D MR spectroscopy in detecting, localizing, and estimating the volume of initial primary prostate cancer as compared to the current standard work-up using TRUS-guided biopsy. All imaging findings will be correlated with "gold standard" step slice histological examination. The hypothesis is that the combination of noninvasive imaging will improve the preoperative work-up as compared to the current approach.
2. To evaluate FCH-PET for the restaging of prostate cancer after biochemical relapse in a large patient cohort. This will run in parallel to the work-up of primary prostate cancer, as the FCH radiopharmaceutical will be available during the time of study at absolutely no cost to patients or CHUV. A number of studies have demonstrated the benefits of F-18-FCH-PET/CT for these patients and this indication is currently not reimbursed by Swiss obligatory health insurance providers.

ELIGIBILITY:
PRIMARY PROSTATE CANCER

Inclusion Criteria:

* Age ≤ 80 years
* Karnofsky index ≥ 80
* First prostate biopsy
* Presence of at least one of the following:

  * Total PSA 10 ng/mL
  * Total PSA 2.5-10 ng/mL with free-PSA <20% and/or PSA velocity 0.75 ng/mL/year
  * Suspicious hypoechoic lesion at TRUS and/or suspicious finding at digital rec¬tal examination
* Informed signed consent.

Exclusion Criteria:

* Impaired capacity to consent
* Coexistence of clinically-proven prostate cancer
* Neoadjuvant hormonal treatment (including 5-α reductase inhibitors)
* Contraindications to surgery
* Contraindications to MR Imaging (see below)

PROSTATE CANCER RELAPSE

Inclusion Criteria:

* Age ≤ 90 years
* Karnofsky index ≥ 80
* Previous treatment for prostate cancer
* No clinical recurrence based on standard work-up (abdominal / pelvic CT, MRI, and bone scintigraphy)
* Biochemically proven relapse of prostate cancer (PSA > 0.2 ng/mL after prostatectomy, nadir PSA+2 ng/mL (Phoenix definition) or ≤ 3 successive rising PSA levels (ASTRO definition) after curative radiotherapy).
* Informed signed consent.

Exclusion Criteria:

* Coexistence of another clinically-proven cancer
* Contraindications to surgery or radiation therapy treatment

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary prostate cancer: Patients referred with a suspicion of prostate cancer based on elevated PSA and rectal examination in whom a prostate biopsy is planned and radical prostatectomy is envisioned in the event of a positive biopsy finding
  Prostate cancer relapse: Patients previously treated for prostate cancer and being investigated for biochemical relapse for whom surgical or radiation therapy is envisioned in the event of a positive FCH-PET finding
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of FCH PET/CT, MR imaging, 3-D MR spectroscopy, and fusion PET/MR imaging for the intraprostatic localization of cancer in patients with radical prostatectomy as compared to histology as the gold standard | After prostatectomy (week 7-9 if Gleason score ≥ 8, week 7-15 if Gleason <8)
For prostate cancer patients with relapse: To determine the impact of FCH-PET imaging for localizing relapse patients in patients with biochemical failure as compared to the standard clinical workup | After PET/CT, week 1-2

SECONDARY OUTCOMES:
To determine if imaging allows for a reliable estimation of tumor volume, as these limits imply a significantly different prognosis in elderly patients (insignificant disease = volume <0.5 cm3 vs. significant disease ≥0.5 cm3) | After prostatectomy (week 7-9 if Gleason score ≥ 8, week 7-15 if Gleason <8)
To determine the utility of dynamic PET imaging using 10 × 1 min acquisitions (0-9 min) as compared to a 5 min static acquisition starting 3 min and a delayed static whole-body acquisition (1 hour after radiotracer injection) | During PET/CT, week 1-2
To determine the impact of parametric PET/CT imaging based on dynamic PET acquisi¬tions with kinetic modeling | During PET/CT, week 1-2
Impact of image-guided biopsies in obtaining adequate tissue samples for histological examination as compared to TRUS-guided extended systematic 12-core biopsies | After TRUS biopsies (week 3)
For prostate cancer patients with relapse: To investigate the potential link between the overall accuracy of FCH and the serum androgen profile (total and free testosterone level) at the day of PET acquisition | After PET/CT, week 1-2

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, PhD MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, CH, Switzerland

IPD SHARING:
Plan to Share IPD: No